CLINICAL TRIAL: NCT03388528
Title: Phase II Feasibility Study of the Efficacy and Acceptability of a Low Residue Diet in Adult Patients With Mitochondrial Disease
Brief Title: Low Residue Diet Study in Mitochondrial Disease
Acronym: LRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/NE/0193
Record Dates: First submitted 2017-10-27; First posted 2018-01-03 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-06

CONDITIONS: Mitochondrial Diseases
Keywords: Dysmotility; Microbiome; Transit Time; Gastrointestinal
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Intervention Model Description: Forty patients with a genetically or biochemically proven diagnosis of mitochondrial disease will be recruited from the mitochondrial Clinics for Research and Service in Themed Assessments (CRESTA) clinic and / or Medical Research Council Mitochondrial Disease Patient Cohort Study in Newcastle
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This is a single arm study where forty patients with a genetically or biochemically proven diagnosis of mitochondrial disease will be recruited from the mitochondrial CRESTA clinic and / or Medical Research Council Mitochondrial Disease Patient Cohort Study in Newcastle. All forty patients will be assessed prior to and following a 12 week low residue diet study intervention.
  Interventions: Dietary Supplement: Low Residue Diet Intervention

INTERVENTIONS:
Dietary Supplement: Low Residue Diet Intervention — All patients will be provided with a LRD plan (< 10g fibre per day) for 12 weeks between visits 2 and 3. They will also be supplemented with multivitamin and mineral tablet or liquid (Forceval) to meet nutrient requirements (prescribed as standard care). The dietitian will provide written and oral information about the LRD and weekly telephone calls to assess patient's progress on the diet.

SUMMARY:
Slow movement of patients guts is referred to as intestinal dysmotility, and is increasingly recognised as a debilitating manifestation of mitochondrial disease both in adults and children.

To date, symptoms of slow gut movements have been managed with laxatives and drugs that increase movement of the guts with variable results. A low residue diet is a form of low fibre diet (<10g fibre per day) that is used to minimise symptoms of poor movement of the guts. This reduces fecal volume and bulk, and hence gut workload, ensuring limited bowel activity and colonic rest. It has been shown to be well accepted in other conditions associated with slow gut movements. However, its role in patients with mitochondrial disease is unknown. The investigators are particularly interested in:

* Does a low residue diet (low fibre) cause a change in the number of stools per week and stool consistency?
* Is a low residue diet tolerated well and easy to comply with?
* Does a low residue diet reduce gut symptoms of abdominal pain, bloating, and constipation?
* Does a low residue diet improve quality of life and disease burden?
* Does a low residue diet affect the bacteria in the gut?
* Can we prove by X-ray that movement of food through the gut is slowed in patients with mitochondrial disease, and whether a low residue diet alters the speed of movement of food through the gut?
* Can a low residue diet change patients physical activity levels?
* Does a low reside diet change dietary patterns and food intake?
* Does a low residue diet alter anthropometrics, such as weight, body mass index and waist to hit ratio?
* Can a low residue diet improve kidney and liver function and lipid profile in blood samples?

The investigators hope that by looking at these areas that a low residue diet may be able to improve patients slow gut movements, health, quality of life and disease burden.

DETAILED DESCRIPTION:
Intestinal dysmotility is increasingly recognised as a debilitating manifestation of mitochondrial disease both in adults and children (1). It is a frequent symptom of other neurological conditions including Cerebral Palsy, Multiple Sclerosis and Parkinson's Disease. Symptoms of intestinal dysmotility are often overlooked and frequently under-diagnosed in its early stages.

Indeed, in its most severe form, intestinal dysmotility may manifest as intestinal pseudo obstruction (IPO), characterised by a clinical picture suggestive of mechanical obstruction, exemplifying the need for early detection and management. To date, symptoms of intestinal dysmotility in slow transit time constipation, limited fluid and calorie intake, weight loss, and small intestinal bacterial overgrowth and in severe cases intestinal pseudo obstruction (2, 3). Moreover, the bacteria that reside within the gastrointestinal (GI) tract compete for nutrients, contributing to weight loss due to malabsorption of fat (4), protein and carbohydrates (5, 6), vitamin (7-11) and iron deficiency (12) are often evident. Further problems include poor digestion and absorption food, an impaired immune system, and an impaired drug absorption ability, all of which influence patient health, quality of life and increases National Health Service (NHS) costs.

A low residue diet is a form of low fibre diet (<10g fibre per day) that is used to minimise symptoms of intestinal dysmotility by reducing faecal volume and bulk and hence bowel workload, ensuring limited bowel activity and colonic rest. It has been shown to be both tolerable and efficacious in other conditions associated with intestinal dysmotility; however, its role in patients with mitochondrial disease and intestinal dysmotility, is unknown.

This feasibility study proposes to systematically gather data on whether a low residue diet is tolerable and has an effect on intestinal dysmotility and health-related quality of life in in patients with mitochondrial disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 and over.
* Genetic or biochemical confirmation of mitochondrial disease.
* ROME III criteria of constipation (Appendix 2).
* Stable gastrointestinal drug regimen prior to commencement of study, at least 3 months prior study inclusion.
* No known hypersensitivities to any of the ingredients in the preparations.
* Not already implementing a low residue diet.
* Competent to make such decisions in the opinion of the investigator.
* Females of child bearing age require a negative pregnancy test.

Exclusion Criteria:

* Patients with known allergies to any adjuncts in the dietary preparation
* Patients with bowel obstruction
* Females who are pregnant, lactating or planning a pregnancy.
* Planned surgery during the course of the trial.
* Participation in another drug trial concurrently or in the preceding 12 weeks.
* Any condition which would put the participant at risk if they were to take part in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Assess tolerability of a Low Residue Diet (LRD) in mitochondrial patients | Change from baseline to 12 weeks
  Tolerability of the LRD will be assessed using food diaries
Stool Frequency and consistency | Change from baseline to 12 weeks
  Assess stool consistency according to the Bristol Stool Form scale. Patients will select from the following to describe their stool consistency:
  Type 1: Separate hard lumps, like nuts Type 2: Sausage-like but lumpy Type 3: Like a sausage but with cracks in the surface Type 4: Like a sausage or snake, smooth and soft Type 5: Soft blobs with clear-cut edges Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces

SECONDARY OUTCOMES:
Gastrointestinal Dysmotility | Change from baseline to 12 weeks
  To determine the impact of a LRD on GI dysmotility symptoms using Assessment of Constipation-Symptom (PAC-SYM) questionnaire.
Disease Burden | Change from baseline to 12 weeks
  To determine the effect of LRD on patients Disease burden as assessed by the Newcastle Mitochondrial Disease Adult Scale (NMDAS) disease burden and quality of life. This is a questionnaire developed and validated by Wellcome Centre for Mitochondrial Research, Newcastle upon Tyne. This is a scored questionnaire that encompasses questions on patient's disease burden encompassing:
  Current Function: Vision with usual glasses or contact lenses; Migraine Headaches; Seizures; Stroke like episodes; Encephalopathic Episodes; Gastro-intestinal symptoms; Diabetes mellitus; Respiratory muscle weakness and Cardiovascular system.
  Current Clinical Assessment: Visual acuity; Ptosis; Chronic Progressive External Ophthalmoplegia; Dysphonia/Dysarthria; Myopathy; Cerebellar ataxia; Neuropathy; Pyramidal Involvement; Extrapyramidal and Cogitation.
  These are all included under the NMDAS questionnaire and are used by clinical care teams to help determine patient's current disease burden.
Gut Microbiome changes | Change from baseline to 12 weeks
  Assess effect of a LRD on gut metagenomics
Gut Microbiome Comparison | Baseline only (prior to any intervention)
  A comparison of the gut microbiome composition and diversity assessed by sequencing, between healthy controls and mitochondrial patients prior to the LRD intervention.
Food Intake | Change from baseline to 12 weeks
  To assess the impact of a LRD on food intake (Food Frequency Questionnaire (FFQ) will be completed for 72 hours (1 day over the weekend and 2 days during the week).
Colonic Transit Time | Change from baseline to 12 weeks
  Colonic transit time (CTT) as assessed by plain abdominal X-ray following ingestion of oral colonic marker ingestion.
Physical Activity | Change from baseline to 12 weeks
  Activity level (GeneActiv 7-10 days).
Biochemistry | Change from baseline to 12 weeks
  The Biochemistry department in the Royal Victoria Infirmary in Newcastle upon Tyne will be provided with whole blood. Using this they will measures liver enzymes (alanine transaminase, aspartate aminotransferase, gamma-glutamyl transpeptide), alkaline phosphatase, albumin, bilirubin, lipid profile and C-Peptide tests.
Gastrointestinal Health | Change from baseline to 12 weeks
  To determine the impact of a LRD on patient GI symptoms using the Gastrointestinal Quality-of-Life Index. This includes defecation characteristics including laxative use and reported abdominal symptoms categorized as pain or cramps and bloating or flatulence according to five classifications (1, none; 2, mild; 3, moderate; 4, severe; or 5, very severe).
Anthropometrics | Change from baseline to 12 weeks
  Weight (kg)
Physical Measurements | Change from baseline to 12 weeks
  Body Mass Index
Physical Dimensions | Change from baseline to 12 weeks
  Waist to hip ratio (inches)
Haematology | Change from baseline to 12 weeks
  The Haematology department in the Royal Victoria Infirmary in Newcastle upon Tyne will be provided with whole blood. Using this they will provide a Full blood count, Haematocrit screen, Ferritin, Vitamin B12, HbA1c and Folate.

CONTACTS AND LOCATIONS:
Overall Officials: Grainne S Gorman, MD, Principal Investigator — Newcastle University
Locations (1):
- Grainne Gorman, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Patients will be anonymised, and only raw outcome data will be shared in conjunction with collaborators of the Wellcome Centre for Mitochondrial Research .

REFERENCES:
- [Derived] Houghton D, Ng YS, Jackson MA, Stefanetti R, Hynd P, Mac Aogain M, Stewart CJ, Lamb CA, Bright A, Feeney C, Newman J, Turnbull DM, McFarland R, Blain AP, Gorman GS. Phase II Feasibility Study of the Efficacy, Tolerability, and Impact on the Gut Microbiome of a Low-Residue (Fiber) Diet in Adult Patients With Mitochondrial Disease. Gastro Hep Adv. 2022 Jul 1;1(4):666-677. doi: 10.1016/j.gastha.2022.03.007. eCollection 2022. PMID 39132075